CLINICAL TRIAL: NCT06966908
Title: Hospital-Based Management of Patients With Chronic Hepatitis B Virus Infection
Status: Enrolling by invitation | Type: Observational
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Liang Peng, Professor, Third Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: PL19
Record Dates: First submitted 2025-04-18; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; linkage to care; management
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HBsAg-positive patients in non-hepatology/non-infectious disease departments
  Interventions: Other: Facilitate the referral of in-hospital chronic hepatitis B patients and provide treatment and follow-up in the infectious disease department.

INTERVENTIONS:
Other: Facilitate the referral of in-hospital chronic hepatitis B patients and provide treatment and follow-up in the infectious disease department. — After visiting the hospital, high-risk HBV patients are prescribed HBsAg testing by their primary physician. If HBsAg positivity is detected in patients from non-infectious disease departments, their lab reports will include a reminder to visit the Hepatitis B Health Clinic. Some primary physicians may also request an infectious disease consultation or recommend patient referral. Additionally, within two weeks, the Hepatitis B Specialist Assistant will contact the patients by phone to provide referral recommendations. Once referred to the Hepatitis B Health Clinic, physicians will conduct health education, complete liver function and virological assessments, and develop individualized treatment and follow-up plans.

SUMMARY:
Starting in 2022, the Third Affiliated Hospital of Sun Yat-sen University implemented the "Hot Wave Project," an integrated HBV infection prevention and control system encompassing patient education, screening, referral, treatment, and follow-up. This system is now being expanded to the Sixth Affiliated Hospital and Fifth Affiliated Hospital of Sun Yat-sen University. Additionally, a multicenter, in-hospital cohort study on HBV management has been initiated.The primary aim of this study is to increase the referral rate from to 50% for HBsAg-positive patients from non-hepatology/non-infectious disease departments. The secondary objective is to improve the treatment rates of HBV-infected individuals in non-hepatology/non-infectious disease departments, especially the population diagnosed but untreated (DBU). Additionally, the study seeks to analyze the cost-effectiveness and clinical benefits of the in-hospital HBV screening and management strategy.

DETAILED DESCRIPTION:
The "Hot wave Project" aims to establish a multicenter management cohort for HBsAg-positive patients within hospitals. Led by infectious disease specialists, the program conducts regular hepatitis B training sessions for hospital staff to enhance their understanding of HBV prevention and control. This initiative seeks to increase HBsAg screening rates overall and encourage patients from non-infectious disease departments to seek referrals to specialized care.

For all paper reports containing HBsAg test results, a remark is added stating: "HBsAg (+) - Recommended to visit the Hepatitis B Health Clinic in the Infectious Disease Department." Positive HBsAg results are automatically extracted by the information system and sent to a dedicated computer in the Hepatitis B Health Clinic, enabling centralized digital patient management.

Additionally, the Infectious Disease Department appoints a "Hepatitis B Specialist Assistant" responsible for reviewing HBsAg screening results, notifying HBsAg-positive patients or their attending physicians, and establishing follow-up records for all patients. A "Hepatitis B Health Clinic" is also set up within the department, managed by a specialized medical team that handles the diagnosis, treatment, and education for referred chronic hepatitis B patients.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg-positive patients attending non-infectious disease/hepatology departments at three study centers between January 2025 and December 2025.

Exclusion Criteria:

* HBsAg-positive patients already under regular follow-up in infectious disease/hepatology clinics.
* Chronic HBV patients on regular antiviral treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HBsAg-positive patients attending non-infectious disease/hepatology departments.
Sampling Method: Non-Probability Sample
Enrollment: 16000 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Referral rate | 2 weeks
  Referral rate of HBsAg-positive patients in non-infectious disease departments = Number of HBsAg-positive patients referred to infectious disease departments / Total number of HBsAg-positive patients in non-infectious disease departments.

SECONDARY OUTCOMES:
Antiviral treatment rate | 2 weeks
  Antiviral treatment rate of HBsAg-positive patients in non-infectious disease departments = Number of patients from non-infectious disease departments starting antiviral treatment / Total number of HBsAg-positive patients in non-infectious disease departments.
The cost-effectiveness of in-hospital HBV screening and management strategies | 5 years
  Develop an economic analysis model to explore the cost-effectiveness of in-hospital HBV screening and management strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Liang Peng, Principal Investigator — Third Affiliated Hospital, Sun Yat-Sen University; Zhongsi Hong, Principal Investigator — Fifth Affiliated Hospital, Sun Yat-Sen University; Fangfang Wei, Principal Investigator — Sixth Affiliated Hospital, Sun Yat-sen University
Locations (3):
- China (3):
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided